CLINICAL TRIAL: NCT00553111
Title: Video Tool to Promote Knowledge of Syphilis as Facilitator of HIV Transmission
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jacobi Medical Center (Other)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: 06-09390
Record Dates: First submitted 2007-11-02; First posted 2007-11-05 (Estimated); Last update posted 2007-11-05 (Estimated); Status verified 2007-11

CONDITIONS: Syphilis
Keywords: syphilis; video education; knowledge; black; hispanic
MeSH Terms: conditions — Syphilis

STUDY DESIGN:
Who Masked: Investigator

ARMS (4):
- 1 (Experimental): pre survey, intervention, post test survey
  Interventions: Other: educational video
- 2 (No Intervention): pre test survey and post test survey
- 3 (Experimental): video intervention and post test survey
  Interventions: Other: educational video
- 4 (No Intervention): post test survey

INTERVENTIONS:
Other: educational video — educational video
  Arms: 1; 3

SUMMARY:
During the winter of 2007, the Syphilis Advisory Group and Bureau of STD Control of the NYC Department of Health funded the Emergency Department of Jacobi Medical Center to further evaluate the effectiveness of the Syphilis and Men video in additional settings where men access STD related information and testing and where high-risk groups, such as MSM, frequent. The video was evaluated for promoting knowledge of syphilis, especially as facilitator of HIV transmission, and in encouraging concurrent testing (syphilis and HIV) among men recruited from a community-based organization, an ambulatory care setting, and a dance club.

DETAILED DESCRIPTION:
The Solomon-four group design was applied to assess the effectiveness of the video in raising syphilis knowledge among participants, while controlling for the influence of the pre-test knowledge survey in skewing post-knowledge survey scores. Participants in Group 1 received a pre-test survey, the video intervention, and the post-test survey; Group 2 received the pre-test and post-test surveys; Group 3 received the video intervention and post-test survey; and Group 4 received the post-test survey only. A computer-generated randomization list was used to assign participants to one of the four groups.

ELIGIBILITY:
Inclusion Criteria:

* must speak english or spanish

Exclusion Criteria:

* excluded if hearing or visually impaired

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2006-11; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
The primary outcome was the score on a 10-question measure designed to assess knowledge attained from the syphilis educational video | 20 minutes

SECONDARY OUTCOMES:
A secondary outcome was the decision to be tested for syphilis and HIV | 20 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Chinazo Cunningham, MD, Principal Investigator — Montefiore Medical Center; John Sanchez, MD, MPH, Principal Investigator — Montefiore Medical Center
Locations (2):
- United States (2):
  - New York University Ambulatory Care Pavilion, Manhattan, New York
  - Gay Men of African Descent, Manhattan, New York